CLINICAL TRIAL: NCT05802914
Title: Efficacy of Soft Active Back Exosuit to Reduce the Risk of Occupational Low Back Pain and Injuries
Brief Title: Soft Active Back Exosuit to Reduce Workplace Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyss Institute at Harvard University (Other)
Collaborators: Boston University (Other); Liberty Mutual (Industry); Verve Motion (Unknown); University of Delaware (Other); Industrial Partner (Unknown); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, David Adam Quirk, Principal Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB22-0308; 4UH3AR076731-02 (NIH)
Record Dates: First submitted 2023-03-02; First posted 2023-04-07 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain; Musculoskeletal Pain; Low Back Injury
Keywords: Exoskeleton; Ergonomics; Wearable Robotics; Exosuit; Occupational Injury
MeSH Terms: conditions — Low Back Pain; Musculoskeletal Pain; Occupational Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into an exosuit or a control group using a 2:1 stratified ratio. Strata will be developed based on workplace, lifetime back pain history, and job tenure (>90 days). Participants in each group will complete regular workplace tasks while wearing or not wearing a back exosuit respectively.
Who Masked: Outcomes Assessor
Masking Description: Because of the transparency of a back exosuit, it is not feasible to blind participants and study team members. However, an independent blind statistician will perform our primary intention to treat analysis on our primary outcome measures. The statistician will perform analysis consistent with our statistical analysis plan, transforming data prior to knowledge of group assignment.
  Additional secondary analysis will be performed on open labeled data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Exosuit (Experimental): Exosuit refers to a soft active back exosuit. Participants in the exosuit arm will be fitted to a personal back exosuit device. Participants will be trained on how to use the device (retrieval, donning, powering up, mode switching, and doffing). Participants will be instructed to use the device at work, emphasizing they wear it whenever it seems practical (e.g. lifting) for as long as it remains comfortable. Associates from Verve Motion will check in with exosuit participants to address comfort issues and help participants integrate the exosuit into their workday.
  Interventions: Device: Back Exosuit
- Control (No Intervention): Control participants will not be assigned a back exosuit. Participants in the control group will perform workplace tasks as normal, completing study surveys at baseline and monthly for 4 months that are identical to exosuit group.

INTERVENTIONS:
Device: Back Exosuit — The back exosuit is a soft wearable robotic suit designed to improve a wearer physiology, kinetics, kinematics to reduce the possibility of injury. The back exosuit is primarily composed of textiles that wrap around an individual's shoulder (backpack) and thighs (thigh wrap) to serve as anchor points. An actuating element attaches to those anchor elements to provide assistive forces while the user performs a physical activity. The soft wearable robot integrates sensing components to be able to detect user biomechanics and device function and actuating elements via algorithms that command the actuation based on users' intent. To encourage usability, the device is easy to don and intuitive to use. This back exosuit has demonstrated significant reductions in back (18%), hip (11%) and knee (22%) extensor muscle activity during a 1-hour workplace simulation task when compared to lifting without a suit.
  Other Names: Verve SafeLift Suit
  Arms: Exosuit

SUMMARY:
The goal of this clinical trial is to determine if a wearable back exosuit can make it safer and easier for workers who bend, lift, and lower objects in an industrial setting.

Many studies have shown that wearable back exoskeletons or exosuits can provide helpful forces making a person's back muscles work less. It is believed that exosuits can lower a person's level of workplace effort and fatigue, making it less likely for them to have back pain at work. Back exosuits could be a solution to make a job easier, but how well they work in the real-world over a long period of time is unclear.

The investigators want to know if workers who wear a back exosuit during the workday will have lower rates of lower back pain or injury than those who are not wearing a back exosuit. The investigators also want to know how well exosuit technology integrates into the workplace (for example, how this technology improves or hinders job performance).

Participants will be randomized into an exosuit group or control group. Participants in the exosuit group will be given a back exosuit that they can use as much as they want at work. All participants will complete surveys monthly.

Researchers will compare the exosuit group to the control group to see if using a back exosuit in a workplace can reduce a person's risk and impact of low back injury or pain. The investigators also want to see if a back exosuit impacts job productivity and if participants find the exosuit becomes useful or bothersome over time.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Works as a full-time (>35 hours/ week) employee for our Industrial Partner
* Regularly bends, lifts, or lowers objects below hip height >50% of their working day for multiple periods lasting more than 1 hour without sitting
* Can read and speak in English
* Has internet access
* Has completed an Exosuit Shift Demonstration
* Thigh circumference is > 19" and < 32"
* Back length (Neck to Iliac Crest) is >18"

Exclusion Criteria:

* Temporary workers not directly employed by our Industrial Partner
* Diagnosed or self-reported sensory motor disorders (stroke, Parkinson's disease, ALS, multiple sclerosis, spinal cord injury, etc.)
* Use of a pacemaker or other powered, implanted medical devices
* Medical condition that would make the participant likely to break bones (i.e., osteoporosis or osteopenia)
* Spinal fracture in the past 2 years
* Spinal surgery at multiple vertebral levels in the participant's lifetime, including vertebroplasty but excluding injections, such as steroids, nerve blockers, etc.
* Sought medical care for spinal surgery at a single vertebral level in the past 2 years, including vertebroplasty but excluding injections, such as steroids, nerve blockers, etc.
* Current malignant cancer
* Currently pregnant
* Skin issues / sensitivity that an exosuit could exacerbate (e.g., thin skin, sensitive skin, easy rashing, easy bruising or skin conditions, Epidermolysis Bullosa, etc.)
* A current episode of upper back or neck pain, requiring modified duties at work
* A recent episode of LBP resulting in pain (sharp, shooting, burning), radiating below one or both legs (past mid-thigh) in the last 3 months (e.g., sciatica)
* A recent episode of back pain resulting in time off work, modified duties, or seeking medical attention in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-04-26 (Actual); Study Completion 2025-04-26 (Actual)

PRIMARY OUTCOMES:
Level of work-interfering low back pain (changes over time and differences between groups) | Baseline, Months (1-4)
  The Cornell Musculoskeletal Discomfort Questionnaire (MDQ) is a composite score that considers the frequency, severity, and work interference of body aches and pains. The back pain score will be evaluated between the 2 groups at 5 time points.
Self-reported incidence of low back pain (changes over time and differences between groups) | Baseline, Months (1-4)
  The definition of low back pain highly influences incidence rates. Low back pain incidence will be identified as a meaningful change (answering in the affirmative with a previous negative response) to the following self-report measures:
  Reporting a Cornell MDQ low back pain score >13.5 Answering yes to: "In the past month, have you felt low back pain that caused you to change your activities for at least 3 days (i.e., have you noticed avoiding certain movements or moving differently than you normally do)?" Answering yes to: "In the past month, have you seen a health care provider for low back pain (i.e., a doctor, nurse, physical therapist, chiropractor, or another health care provider)?" Answering yes to: "In the past month, have you taken time off work for low back pain?"
Workplace reported incidence of a low back injury (differences between groups) | Continuously from randomization to 4 months
  Our industrial partner will record if a participant reports a workplace low back injury. The rates of reported events will be measured in each group.

SECONDARY OUTCOMES:
Self-reported severity of low back pain (changes over time and differences between groups) | Baseline, Months (1-4)
  Back pain severity refers to the level of intensity and the occupational or medical consequence of back pain. The following self-report measures will determine these values.
  Intensity:
  Numerical rating scale of back pain (average and worse imaginable)
  Medical consequence:
  Frequency of using over the counter and prescription medication for LBP Frequency of seeing various types of medical providers for LBP
  Occupational Consequences:
  Number of days off following LBP Number of days on modified work duties following LBP
Workplace reported severity of low back pain (differences between groups) | Continuously from randomization to 4 months
  Our industrial partner will record the severity of a low back injury (LBI) in the following ways:
  Number of insurance claims for LBI Number of days off work following a LBI Number of days of reduced work productivity (days on modified duties) following a LBI Medical payouts for LBI claims
Self-reported intensity of global pain (changes over time and differences between groups) | Baseline, Months (1-4)
  Beyond low back pain participants will report on total body discomfort and the intensity of discomfort at various joints:
  Total body discomfort and interference will be evaluated using the Pain, Enjoyment of Lift and General Activity (PEG) 3 Scale.
Self-reported intensity of localized body discomfort (changes over time and differences between groups) | Baseline, Months (1-4)
  The Cornell MSD scale (reference in outcome 1) will also be evaluated at every other body part (for example, ankles, knees, hip, upper back, neck, shoulders, elbows, and wrists).
Self-reported perception of physical fatigue and effort (changes over time and differences between groups) | Baseline, Months (1-4)
  A modified BORG CR-10 scale has been developed with questions focusing on:
  Perceived level of back exertion Perceived level of total body exertion Perceived level of workplace fatigue

OTHER OUTCOMES:
Perceived intervention satisfaction, job productivity, device usability, and device adverse events (changes over time and differences between groups) | Baseline, Months (1-4)
  Various 5 point Likert scales have been developed to probe how a participants relationship with the exosuit and study change over time across the following themes: satisfaction with group assignment, productivity, ability to lift safer, ease to complete work tasks, work satisfaction, support from company, thought of exosuit being a good idea, desire to use an exosuit, ease of using the device, ease of putting on the device, ability to adjust the device, likelihood of experiencing a back injury, levels of fatigue, low back discomfort, feeling the exosuit makes a job too complex, exosuit interference with job time, device comfort, number of times a user must take-off the exosuit during the workday, thermal discomfort, notice of skin issues, uncomfortable skin pressure, bumping or catching objects, experience of balance difficulties, experience of movement restriction

CONTACTS AND LOCATIONS:
Locations (1):
- Undisclosed Location, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study are part of the National Institutes of Health (NIH) Helping to End Addiction Long-term (HEAL) Initiative. As part of the Back Pain Consortium (BACPAC) data form this study will be submitted to the Data Integration, Algorithm Development and Operations Management Center (DAC) following study completion. Researchers will have the possibility to request data from the DAC.
Time Frame: Data will be uploaded to the DAC approximately 6 months to 1 year at study completion. Data may be stored in the DAC indefinitely.
Access Criteria: Formal approval from the BACPAC DAC.

REFERENCES:
- [Background] Quirk DA, Chung J, Schiller G, Cherin JM, Arens P, Sherman DA, Zeligson ER, Dalton DM, Awad LN, Walsh CJ. Reducing Back Exertion and Improving Confidence of Individuals with Low Back Pain with a Back Exosuit: A Feasibility Study for Use in BACPAC. Pain Med. 2023 Aug 4;24(Suppl 1):S175-S186. doi: 10.1093/pm/pnad003. PMID 36794907
- [Background] Zelik KE, Nurse CA, Schall MC Jr, Sesek RF, Marino MC, Gallagher S. An ergonomic assessment tool for evaluating the effect of back exoskeletons on injury risk. Appl Ergon. 2022 Feb;99:103619. doi: 10.1016/j.apergo.2021.103619. Epub 2021 Nov 2. PMID 34740072
- [Background] Hedge A, Morimoto S, McCrobie D. Effects of keyboard tray geometry on upper body posture and comfort. Ergonomics. 1999 Oct;42(10):1333-49. doi: 10.1080/001401399184983. PMID 10582503
- [Background] Baldassarre A, Lulli LG, Cavallo F, Fiorini L, Mariniello A, Mucci N, Arcangeli G. Industrial exoskeletons from bench to field: Human-machine interface and user experience in occupational settings and tasks. Front Public Health. 2022 Nov 21;10:1039680. doi: 10.3389/fpubh.2022.1039680. eCollection 2022. PMID 36478728

DOCUMENTS (1):
  • Informed Consent Form (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT05802914/ICF_000.pdf